CLINICAL TRIAL: NCT06502119
Title: Knowledge, Attitudes, and Practices of Operative Vaginal Birth Among Obstetric Providers in Egypt
Status: Completed | Type: Observational
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Muhamed Ahmed Abdelmoaty Muhamed Alhagrasy, lecturer and consultant at Obstetrics and Gynecology Department., Al-Azhar University
Other Study IDs: Gyne 2024
Record Dates: First submitted 2024-06-27; First posted 2024-07-16 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-07

CONDITIONS: Birth Outcome, Adverse
Keywords: Operative Forceps; Vaginal birth; Birth injuries
MeSH Terms: conditions — Pregnancy Complications; Birth Injuries

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Health Provider: The study will include obstetricians and gynecologists practicing in Egypt. These healthcare professionals specialize in the management of pregnancy, childbirth, and women's reproductive health. Participants will be recruited from various healthcare settings, including public and private hospitals, ensuring a diverse representation of clinical experiences and perspectives on operative vaginal birth practices. All participants must actively engage in obstetric care and possess direct experience with operative vaginal births, allowing for an in-depth exploration of their knowledge, attitudes, and practices related to this procedure within the Egyptian healthcare context.
  Interventions: Other: Designed Questionnaire

INTERVENTIONS:
Other: Designed Questionnaire — Participants in this study, comprised solely of obstetricians and gynecologists practicing in Egypt, will complete a self-administered questionnaire designed to assess their knowledge, attitudes, and practices related to operative vaginal birth. The questionnaire includes four sections: the first gathers demographic data such as name, gender, and years of experience in childbirth care; the second focuses on participants' practices regarding the frequency and types of operative vaginal birth used (forceps, ventouse) and reasons for their use; the third evaluates knowledge of outcomes associated with operative vaginal birth through multiple-choice questions; and the fourth explores attitudes towards operative vaginal birth, including opinions on hospital rates and policy appropriateness. Completion and return of the questionnaire, which takes approximately 5 to 10 minutes, will be considered as consent to participate in the study.

SUMMARY:
The goal of this observational study is to evaluate the knowledge, attitudes, and practices of operative vaginal birth among obstetric providers in Egypt. The main questions it aims to answer are:

* What is the level of knowledge among obstetric providers regarding operative vaginal birth?
* What are the attitudes and practices of obstetric providers towards operative vaginal birth?

Participants will:

* Complete a detailed questionnaire assessing their knowledge, attitudes, and practices related to operative vaginal birth.
* Provide demographic information to contextualize their responses.

ELIGIBILITY:
Inclusion Criteria:

* Licensed Obstetricians: Only obstetricians who are currently licensed to practice in Egypt.
* Active Practice: Obstetricians who are actively practicing in hospitals or clinics in Egypt.
* Experience: Obstetricians with a minimum of one year of experience in obstetrics and gynecology.
* Consent: Willingness to participate and provide informed consent.
* Language: Ability to understand and complete the questionnaire in English.

Exclusion Criteria:

* Non-Obstetricians: Healthcare providers who are not obstetricians.
* Inactive Practice: Obstetricians who are not currently practicing in Egypt.
* Insufficient Experience: Obstetricians with less than one year of experience in the field.
* Non-Consent: Individuals who do not provide informed consent to participate in the study.
* Language Barrier: Obstetricians who are unable to understand and complete the questionnaire in English.

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: This study focuses exclusively on obstetricians and gynecologists practicing in Egypt. These healthcare professionals are actively involved in providing obstetric care and have direct experience with operative vaginal births. Participants will be recruited from various healthcare settings, including public and private hospitals, ensuring a diverse representation of clinical perspectives and experiences across different practice environments within Egypt.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2024-07-20 (Actual); Primary Completion 2025-06-01 (Actual); Study Completion 2025-06-01 (Actual)

PRIMARY OUTCOMES:
Knowledge of Operative Vaginal Birth Among Obstetric Providers | Within 6 months of study commencement.
  The level of knowledge regarding operative vaginal birth among obstetric providers, assessed using a validated questionnaire. The knowledge score will be based on correct responses to a series of questions about indications, techniques, benefits, and risks associated with operative vaginal birth.
Attitudes Toward Operative Vaginal Birth Among Obstetric Providers | Within 6 months of study commencement.
  The attitudes of obstetric providers towards operative vaginal birth, measured using a Likert scale in the validated questionnaire. Providers will rate their agreement with statements related to their perceptions and opinions on the use of operative vaginal birth.
Practices of Operative Vaginal Birth Among Obstetric Providers | Within 6 months of study commencement.
  The frequency and context of operative vaginal birth practices among obstetric providers, as reported in the validated questionnaire. This measure will include the number of operative vaginal births performed, preferred techniques, and any barriers to performing these procedures.
Rate of Cesarean Sections Among Participants | Within 6 months of study commencement.
  The percentage of Cesarean sections performed by the obstetric providers participating in the study, as reported in the validated questionnaire. This measure aims to correlate knowledge, attitudes, and practices with the actual rate of Cesarean sections.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty od Medicine, Department of Obstetrics and Gynecology., Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
As part of this study, Individual Participant Data (IPD) will be shared to facilitate transparency and enable further research in the field of operative vaginal birth practices among obstetricians and gynecologists in Egypt. De-identified IPD will include demographic information, responses from the questionnaire assessing knowledge, attitudes, and practices related to operative vaginal birth, and any additional data pertinent to the study outcomes. Access to the IPD will be granted to researchers with approved proposals demonstrating scientific merit and ethical approval. Data will be made available through a secure, encrypted transfer mechanism, and all users will be required to sign a Data Use Agreement (DUA) outlining terms for responsible data use and confidentiality.
Supporting Information: Study Protocol, SAP
Time Frame: Data collection for the study will commence on [1, July, 2014] and conclude by [30, October, 2024]. IPD will be accessible for sharing beginning [30, December, 2024] and will remain available for a period of [2 years] following publication of primary study results.
Access Criteria: Access to IPD will be granted to researchers with scientifically sound proposals aimed at advancing knowledge in the field of operative vaginal birth practices among obstetricians and gynecologists in Egypt. Proposals must include evidence of ethical approval from an institutional review board or equivalent ethics committee. Researchers affiliated with recognized academic, medical, or research institutions will be eligible. Access requests will be evaluated based on the scientific merit of the proposal, feasibility of the research aims, and potential contribution to improving health outcomes. All users must sign a Data Use Agreement (DUA) ensuring confidentiality, ethical data use, and prohibiting attempts to re-identify participants.